CLINICAL TRIAL: NCT01293838
Title: Cipralex® for Anxiety Disorders in Adolescents: Clinical and Physiological Changes Associated With Open Label, Flexible-dose Treatment
Brief Title: Cipralex® for Anxiety Disorders in Adolescents
Acronym: CAP-E
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ottawa (Other)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Dr. Martine Flament, MD, PhD, FRCPC, Director of Youth Research Unit, University of Ottawa Institute of Mental Health Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMHR REB#2007036; 123485 (Registry Identifier: Office of Clinical Trials, Health Canada)
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Last update posted 2011-02-11 (Estimated); Status verified 2011-01

CONDITIONS: Anxiety Disorder
Keywords: Adolescents; Anxiety Disorder; Cipralex; Social Phobia; Separation Anxiety Disorder; Panic Disorder; Generalized Anxiety Disorder; physiological arousal; stress response; salivary cortisol; salivary alpha-amylase; heart rate variability
MeSH Terms: conditions — Anxiety Disorders; Phobia, Social; Anxiety, Separation; Panic Disorder; Generalized Anxiety Disorder; Fractures, Stress | interventions — Dexetimide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Cipralex® — Based on a starting rate of 5 mg/day, increased by 5 mg every 2 weeks to a maximum of 20 mg/day for weeks 7-16, each participant will receive up to:
  * 10 mg tablets: 28
  * 20 mg tablets: 84
  Total for 30 participants:
  * 10 mg tablets: 840
  * 20 mg tablets: 2520
  Continuation study for participants who respond to Cipralex - Across 12 weeks, each participant will receive up to:
  *20 mg tablets: 84
  Total for continuation study for all participants (assuming a 60% response rate, N=18):
  *20 mg tablets: 1512
  Other Names: Chemical/Pharmaceutical alternative name: Escitalopram

SUMMARY:
The primary objective is to examine whether Cipralex® is effective and safe in the treatment of anxiety disorders in youth. The secondary objective is to identify changes in arousal and stress response from pre- to post-treatment with Cipralex® in youth with anxiety disorders.

DETAILED DESCRIPTION:
Anxiety disorders are the most common mental illnesses of adolescence, with an overall prevalence ranging from 5.0% to 10.8% (Costello et al, 1996; Ford et al, 2003; Fergusson et al, 1993; Shaffer et al, 1996; Verhulst et al., 1997). Six- to 12-month prevalence has been estimated to be 0.5-2.4% for separation anxiety disorder (SAD), 2.1-4.6% for overanxious disorder (OAD), the DSM-III antecedent of generalized anxiety disorder (GAD), 1.7-6.9% for social phobia (SP), and 0.3-1.2% for panic disorder (PD) (Bowen et al, 1990; Fergusson et al, 1993; Ford et al, 2003; Lewinsohn et al, 1993; Romano et al, 2001; Verhulst et al, 1997). In the US National Comorbidity Survey, the median age of onset for anxiety disorders was 11 years (range 6-21 years), which was much younger than for substance use disorders (20 years) and mood disorders (30 years) (Kessler, 2005). However, anxious youth often go undiagnosed and untreated, possibly because they tend to be compliant and nondisruptive (Esser et al, 1990). This is of concern since research suggests that youth with untreated anxiety disorders are more likely to develop significant problems later in life, such as continued anxiety, depression, substance abuse, suicide attempts, educational underachievement, and impaired psychosocial functioning (Pine et al, 1998; Woodward & Fergusson, 2001).

The existing literature on pharmacological treatment of anxiety disorders in adolescents is limited, but suggests that the selective serotonin reuptake inhibitors (SSRIs) are the treatment of choice for pervasive and impairing anxiety disorders in youth (Reinblatt & Walkup, 2005). A few randomized controlled trials (RCT) provide support for the use of SSRIs such as fluvoxamine and fluoxetine for the treatment of SAD, GAD and SP. Cipralex® is a newer SSRI whose use for treatment of anxiety disorders in adolescents has been documented in only one previous open trial (Isolan et al., 2007). Results from this study and a few RCTs conducted in adults with anxiety disorders suggest that Cipralex® should be effective and safe for relieving symptoms of anxiety in adolescents.

Primary objectives: (1) to assess the clinical and psychosocial changes associated with 16-week open-label treatment with Cipralex® (10 to 20 mg/day) in adolescents with SAD, SP, PD and/or GAD; (2) to assess the tolerance and safety of Cipralex® (10 to 20 mg/day for 16 weeks) in adolescents with SAD, SP, PD and/or GAD.

Secondary objective: (1) to investigate changes in physiological measures of arousal and stress response (i.e., heart rate variability, salivary concentrations of cortisol and alpha-amylase, acoustic startle response,) using standardized laboratory stressors, before and after treatment with Cipralex® (10 to 20 mg/day for 16 weeks) in youth with anxiety disorders.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of (1 or more)
* Social Phobia
* Generalized Anxiety Disorder
* Separation Anxiety Disorder
* Panic Disorder
* Comorbid depression allowed

Exclusion Criteria:

* Unstable medical condition
* Substance use disorder
* Current diagnosis of OCD
* Lifetime diagnosis of developmental delay, pervasive developmental disorder, psychosis

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-03; Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Treatment Efficacy | At week 16
  Measures used to assess treatment efficacy:
  * The Anxiety Disorders Interview Schedule for DSM-IV, Research and Lifetime Version for Children and Parents (Silverman & Albano, 1996)
  * Multidimensional Anxiety Scale for Children (March et al., 1997)
  * Youth Quality of Life Scale (Topolski et al., 2001),
  * Pediatric Anxiety Rating Scale (RUPP, 2002)
  * Beck Depression Inventory-2 (Beck et al., 1996
  * Behavioral and Emotional Rating Scale-2 (Epstein & Sharma, 2004),
  * Clinical Global Impression Scale-Severity and Improvement (Guy, W. & ECDEU, 1976)

SECONDARY OUTCOMES:
Physiological response to stress | At week 18 - see below
  * Trier Social Stress Task for Children (TSST-C)[Baseline and week 18]
  * Salivary cortisol[For baseline, samples will be collected in the home upon awakening/8 am, +30, +60 min, at 4 pm, and at 8 pm on 2 consecutive weekdays. Cortisol will also be measured from samples collected before and after the TSST-C(-1, +10, +20, +30, +45, and +60 min)]
  * Salivary alpha-amylase[Before (-1), and +1, +10, +20, and +30 min after the TSST-C]
  * Heart rate variability[Baseline and during the TSST-C]
  * Acoustic Startle Response[Baseline and in a "fear-potentiated" condition with an ASR system]
  * Urine drug test
Suicide risk | Each treatment visit (baseline then weeks 2, 4, 6, 8, 12, 16, 28)
  At each treatment visit, the clinician will elicit AEs and SAEs, and complete the Columbia-Suicide Severity Rating Scale (C-SSRS) (Posner et al, 2007)

CONTACTS AND LOCATIONS:
Overall Officials: Martine Flament, MD, Principal Investigator — University of Ottawa
Locations (1):
- The University of Ottawa Institute of Mental Health Research, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Posner K, Melvin GA, Stanley B, Oquendo MA, Gould M. Factors in the assessment of suicidality in youth. CNS Spectr. 2007 Feb;12(2):156-62. doi: 10.1017/s1092852900020678. PMID 17277716
- [Background] Costello EJ, Angold A, Burns BJ, Stangl DK, Tweed DL, Erkanli A, Worthman CM. The Great Smoky Mountains Study of Youth. Goals, design, methods, and the prevalence of DSM-III-R disorders. Arch Gen Psychiatry. 1996 Dec;53(12):1129-36. doi: 10.1001/archpsyc.1996.01830120067012. PMID 8956679
- [Background] Fergusson DM, Horwood LJ, Lynskey MT. Prevalence and comorbidity of DSM-III-R diagnoses in a birth cohort of 15 year olds. J Am Acad Child Adolesc Psychiatry. 1993 Nov;32(6):1127-34. doi: 10.1097/00004583-199311000-00004. PMID 8282656
- [Background] Shaffer D, Fisher P, Dulcan MK, Davies M, Piacentini J, Schwab-Stone ME, Lahey BB, Bourdon K, Jensen PS, Bird HR, Canino G, Regier DA. The NIMH Diagnostic Interview Schedule for Children Version 2.3 (DISC-2.3): description, acceptability, prevalence rates, and performance in the MECA Study. Methods for the Epidemiology of Child and Adolescent Mental Disorders Study. J Am Acad Child Adolesc Psychiatry. 1996 Jul;35(7):865-77. doi: 10.1097/00004583-199607000-00012. PMID 8768346
- [Background] Verhulst FC, van der Ende J, Ferdinand RF, Kasius MC. The prevalence of DSM-III-R diagnoses in a national sample of Dutch adolescents. Arch Gen Psychiatry. 1997 Apr;54(4):329-36. doi: 10.1001/archpsyc.1997.01830160049008. PMID 9107149
- [Background] Bowen RC, Offord DR, Boyle MH. The prevalence of overanxious disorder and separation anxiety disorder: results from the Ontario Child Health Study. J Am Acad Child Adolesc Psychiatry. 1990 Sep;29(5):753-8. doi: 10.1097/00004583-199009000-00013. PMID 2228929
- [Background] Lewinsohn PM, Hops H, Roberts RE, Seeley JR, Andrews JA. Adolescent psychopathology: I. Prevalence and incidence of depression and other DSM-III-R disorders in high school students. J Abnorm Psychol. 1993 Feb;102(1):133-44. doi: 10.1037//0021-843x.102.1.133. PMID 8436689
- [Background] Romano E, Tremblay RE, Vitaro F, Zoccolillo M, Pagani L. Prevalence of psychiatric diagnoses and the role of perceived impairment: findings from an adolescent community sample. J Child Psychol Psychiatry. 2001 May;42(4):451-61. PMID 11383961
- [Background] Kessler RC, Berglund P, Demler O, Jin R, Merikangas KR, Walters EE. Lifetime prevalence and age-of-onset distributions of DSM-IV disorders in the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005 Jun;62(6):593-602. doi: 10.1001/archpsyc.62.6.593. PMID 15939837
- [Background] Esser G, Schmidt MH, Woerner W. Epidemiology and course of psychiatric disorders in school-age children--results of a longitudinal study. J Child Psychol Psychiatry. 1990 Jan;31(2):243-63. doi: 10.1111/j.1469-7610.1990.tb01565.x. PMID 2312652
- [Background] Woodward LJ, Fergusson DM. Life course outcomes of young people with anxiety disorders in adolescence. J Am Acad Child Adolesc Psychiatry. 2001 Sep;40(9):1086-93. doi: 10.1097/00004583-200109000-00018. PMID 11556633
- [Background] Reinblatt SP, Walkup JT. Psychopharmacologic treatment of pediatric anxiety disorders. Child Adolesc Psychiatr Clin N Am. 2005 Oct;14(4):877-908, x. doi: 10.1016/j.chc.2005.06.004. PMID 16171707
- [Background] Isolan L, Pheula G, Salum GA Jr, Oswald S, Rohde LA, Manfro GG. An open-label trial of escitalopram in children and adolescents with social anxiety disorder. J Child Adolesc Psychopharmacol. 2007 Dec;17(6):751-60. doi: 10.1089/cap.2007.0007. PMID 18315447
- [Background] March JS, Parker JD, Sullivan K, Stallings P, Conners CK. The Multidimensional Anxiety Scale for Children (MASC): factor structure, reliability, and validity. J Am Acad Child Adolesc Psychiatry. 1997 Apr;36(4):554-65. doi: 10.1097/00004583-199704000-00019. PMID 9100431
- [Background] Topolski TD, Patrick DL, Edwards TC, Huebner CE, Connell FA, Mount KK. Quality of life and health-risk behaviors among adolescents. J Adolesc Health. 2001 Dec;29(6):426-35. doi: 10.1016/s1054-139x(01)00305-6. PMID 11728892
- [Background] Silverman, W. K. & Albano, A. M. (1996). The Anxiety Disorders Interview Schedule for DSM-IV-Child and Parent Versions. San Antonio, TX, Psychological Corporation.
- [Background] Beck, A. T., Steer, R. A., & Brown, G. K. (1996). Manual for the Beck Depression Inventory-2. San Antonio, TX: Psychological Corporation.
- [Background] Epstein, M. H., & Sharma, J. M. (2004). Behavioral and Emotional Rating Scale-2: A strength-based approach to assessment. Austin, TX: PRO-ED.
- [Background] Guy, W. & ECDEU (1976). Assessment Manual for Psychopharmacology. Early Clinical Drug Evaluation Unit.
- [Background] The Pediatric Anxiety Rating Scale (PARS): development and psychometric properties. J Am Acad Child Adolesc Psychiatry. 2002 Sep;41(9):1061-9. doi: 10.1097/00004583-200209000-00006. PMID 12218427
- [Background] Pine DS, Cohen P, Gurley D, Brook J, Ma Y. The risk for early-adulthood anxiety and depressive disorders in adolescents with anxiety and depressive disorders. Arch Gen Psychiatry. 1998 Jan;55(1):56-64. doi: 10.1001/archpsyc.55.1.56. PMID 9435761